CLINICAL TRIAL: NCT00491842
Title: Individuals' Patterns of Disclosure About Huntington's Disease and Association With Adaptation to HD
Brief Title: Individuals Patterns of Disclosure About Huntington s Disease (HD) and the Association With Adaptation to HD
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907179; 07-HG-N179
Record Dates: First submitted 2007-06-23; First posted 2007-06-26 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; Disclosure; Adaptation; Communication; Natural History; Huntington Disease; HD; Phone Interview
MeSH Terms: conditions — Huntington Disease; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- At-risk: Individuals at-risk for HD
- Presymptomatic: Presymptomatic carriers of HD

SUMMARY:
This study will examine the ways in which people reveal their status as a carrier of Huntington s disease (HD) or of being at risk for the disease. It will explore factors that influence decisions about disclosure and how disclosure is made to family members, partners, and close friends.

HD is an inherited, progressive disease. It causes nerve degeneration, motor disturbance, loss of awareness, and psychiatric symptoms. Currently, no effective treatment is available to prevent or delay HD progression. The mean age of onset is 35 to 44 years, and the median survival rate after onset is 15 to 18 years. HD affects about 1 in 10,000 people in the United States, so about 30,000 have HD and more than 200,000 are at risk. Predictive testing for HD has been available since 1993. It can be a life-changing event to learn of being at risk for HD. Disclosure has been studied among people with HD and other diseases, but knowledge about the extent of nondisclosure and disclosure is limited. There is evidence that a person s psychological adaptation to AD may be a factor. Adaptation involves processes that help a person search for meaning in what has happened, attempt to gain control of his or her life, and improve self-esteem in light of the threatening situation.

Participants ages 18 and older who have had a positive genetic test result more than 6 months earlier regarding HD or who have a family history of HD but no predictive testing and who do not have symptoms of HD may be eligible for this study. Recruitment is done through HD clinics, support groups, and online websites and mailing listservs. About 260 people will be in the study. Participants will complete a survey taking 30 to 40 minutes to do. Two survey versions are available: for those who are gene carriers and for those at risk. Participants are asked to complete the version applying to them. The survey can be done online or through a hard copy to complete at home and send to NIH. This survey is anonymous.

Participants will list the adults with whom they have a relationship and up to 10 people they interact with. They will indicate those who know about the HD gene or risk status. They will also list those to whom they have personally made disclosure. The goal is to distinguish if knowing the status or the act of disclosure is more important. Questions also involve discussing the inheritance and features of HD, and participants feelings or concerns about HD gene or risk status. Participants will be asked about their first disclosure experience, most recent experience of it, and timing of disclosure the time between learning of HD status and telling another person about it. There are also questions on decisions of nondisclosure, negative and positive aspects of disclosure for participants, and what health care professionals can do to help participants disclosure decisions.

DETAILED DESCRIPTION:
The proposed study aims to describe presymptomatic and at-risk individuals' patterns of disclosure about Huntington's disease (HD) and HD risk to family and friends, and to investigate whether an association exists between disclosure about HD and psychological adaptation to HD. HD is reported to be one of the conditions most frequently involved in cases of nondisclosure about genetic risk. Little is known about the extent of disclosure and the process of disclosure within the HD population. Evidence suggests that a relationship may exist between disclosure of one's condition to others and psychological adaptation to the condition; however, this theory has never been tested. The conceptual framework of the study is informed by Shelly Taylor's Theory of Cognitive Adaptation. We will use a cross-sectional survey to 1) investigate individuals' patterns of disclosure about HD and 2) assess psychological adaptation to HD. Participants will be recruited from HD clinics, HD support groups, HD websites, and HD online mailing listservs. Eligible participants will be asked to complete either a web-based or a paper survey. The main outcome measure is psychological adaptation to HD.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Men and women who self-report:

  * Testing positive for the HD gene expansion, or
  * Not having undergone predictive genetic testing, but having a grandparent, parent, or sibling who has been clinically diagnosed with HD or has tested positive for the HD gene expansion
* Ability to read and write English

EXCLUSION CRITERIA:

* Children younger than 18
* Manifesting HD symptoms, based on self-report
* Received predictive genetic testing within the past 6 months
* Received predictive genetic test result indicating the absence of the gene expansion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Presymptomatic carriers of HD & Individuals at-risk for HD
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2007-06-22; Primary Completion 2008-03-27 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Social Network Measure Developed Specifically for this Study | Enrollment
  To explore what factors influence decisions about disclosure of HD carrier or risk status in the target population
Social Network Measure Developed Specifically for this Study | Enrollment
  To explore relationships between the three domains of disclosure: to whom individuals are disclosing their HD carrier or risk status, when individuals are disclosing their HD carrier or risk status, and what specific information individuals are disclosing to family members, partners, and close friends.
Social Network Measure Developed Specifically for this Study | Enrollment
  To describe patterns of disclosure in the target population
Psychological Adaptation Scale | Enrollment
  To examine the relationship between individuals patterns of disclosure about HD and HD risk and their psychological adaptation to HD, taking into account other covariates (gender, age, ethnicity, marital status, level of education, known positive gene carrier versus at-risk, and recruitment source).

CONTACTS AND LOCATIONS:
Overall Officials: Lori Erby, Ph.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clarke A, Richards M, Kerzin-Storrar L, Halliday J, Young MA, Simpson SA, Featherstone K, Forrest K, Lucassen A, Morrison PJ, Quarrell OW, Stewart H. Genetic professionals' reports of nondisclosure of genetic risk information within families. Eur J Hum Genet. 2005 May;13(5):556-62. doi: 10.1038/sj.ejhg.5201394. PMID 15770225
- [Background] Craufurd D, Dodge A, Kerzin-Storrar L, Harris R. Uptake of presymptomatic predictive testing for Huntington's disease. Lancet. 1989 Sep 9;2(8663):603-5. doi: 10.1016/s0140-6736(89)90722-8. PMID 2570293
- [Background] Figueiredo MI, Fries E, Ingram KM. The role of disclosure patterns and unsupportive social interactions in the well-being of breast cancer patients. Psychooncology. 2004 Feb;13(2):96-105. doi: 10.1002/pon.717. PMID 14872528